CLINICAL TRIAL: NCT00686192
Title: The Effects of Calcium Supplementation on Adipocyte Metabolism in Overweight Women
Brief Title: Calcium and Lipid Metabolism
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: USDA, Western Human Nutrition Research Center (U.S. Federal Agency)
Collaborators: University of California, Davis (Other); San Francisco General Hospital (Other)
Responsible Party: Janet C. King, PhD, Children's Hospital Oakland Research Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: WHNRC001
Record Dates: First submitted 2008-05-27; First posted 2008-05-29 (Estimated); Last update posted 2008-07-22 (Estimated); Status verified 2008-05

CONDITIONS: Obesity
Keywords: Obesity; Calcium carbonate; Dietary Supplements; Lipolysis
MeSH Terms: conditions — Obesity | interventions — Calcium Carbonate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Dietary Supplement: Calcium Carbonate — 1500 mg per day

SUMMARY:
We hope to determine if supplementing the diet of women who habitually consume low levels of calcium, with 1500 mg of calcium a day for three months will increase fat oxidation and decrease fat storage. We will also measure concentrations of lipids, glucose, hormones and enzymes associated with fat and carbohydrate metabolism to determine alterations and mechanism of the metabolic changes.

DETAILED DESCRIPTION:
The incidence of obesity has rapidly increased in recent years and reached epidemic proportions in the United States. Recent epidemiological data has shown an inverse relationship between calcium intake and body fat and emerging research suggests that inadequate dietary calcium consumption may increase obesity. Studies in mice have shown that an increase in dietary calcium consumption creates a shift in the utilization of energy stores from carbohydrates to fat and a shift in the partitioning of energy from storage (as fat) to expenditure (as heat).

We will give 1500 mg of calcium a day for three months to women who habitually consume low levels of dietary calcium. The following measurements will be made before and after calcium supplementation: body fat by DEXA, lipolysis by infusion of stable isotopes of 1,1,2,3,3-[2H5] glycerol , hepatic glucose production by infusion of stable isotopes of 6,6-[2H2] glucose, lipogenesis by measurement of fatty acid synthase activity (14C radiochemical assay) , mRNA expression ( Real Time Polymerase Chain Reaction) and protein content (ELISA), indirect calorimetry measurement of non-protein respiratory quotient (NPRQ), energy expenditure, fat and carbohydrate oxidation. Serum calcium, glucose, cholesterol, triglycerides, LDL, HDL, parathyroid hormone, leptin, free fatty acids, adiponectin, 1,25(OH)2D, 25(OH)D and urinary calcium excretion will also be measured.

ELIGIBILITY:
Inclusion Criteria:

* BMI between 25 and 30 kg/m2
* Taking oral contraceptives
* Having regular menses

Exclusion Criteria:

* Pregnant
* History of metabolic bone, renal or thyroid disease,
* History of diabetes mellitus, or gestational diabetes mellitus
* Cigarette smoking
* Self-administration of calcium supplements
* Regular aerobic activity, i.e. jogging > 1 mile/day

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2001-09; Primary Completion 2002-07 (Actual); Study Completion 2002-07 (Actual)

PRIMARY OUTCOMES:
Lipolysis by infusion of stable isotopes of 1,1,2,3,3-[2H5] glycerol | 0 and 3 months

SECONDARY OUTCOMES:
Hepatic glucose production by infusion of stable isotopes of 6,6-[2H2] glucose | 0 and 3 months
Lipogenesis by measurement of fatty acid synthase activity (14C radiochemical assay) , mRNA expression ( Real Time Polymerase Chain Reaction) and protein content (ELISA) | 0 and 3 months
Indirect calorimetry measurement of non-protein respiratory quotient (NPRQ), energy expenditure, fat and carbohydrate oxidation | 0 and 3 months
Serum calcium, glucose, cholesterol, triglycerides, LDL, HDL, parathyroid hormone, leptin, free fatty acids, adiponectin, 1,25(OH)2D, 25(OH)D | 0 and 3 months
urinary calcium and sodium excretion | 0 and 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Janet C King, PhD, Principal Investigator — UCSF Benioff Children's Hospital Oakland
Locations (1):
- San Francisco General Hospital, San Francisco, California, United States

REFERENCES:
- See also: USDA Western Human Nutrition Research Center — http://www.ars.usda.gov/main/site_main.htm?modecode=53062500